CLINICAL TRIAL: NCT02358044
Title: A Phase III, Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172/MK-8742 Versus Sofosbuvir/Pegylated Interferon/Ribavirin (PR) in Treatment-Naïve and PR Prior Treatment Failure Subjects With Chronic HCV GT1, 4 or 6 Infection
Brief Title: Efficacy and Safety of Combination Grazoprevir (MK-5172)/Elbasvir (MK-8742) Versus Sofosbuvir + Pegylated Interferon + Ribavirin in Hepatitis C Virus Genotype 1, 4 or 6 Infection (MK-5172-077)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-077; 2014-003836-38 (EudraCT Number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; peginterferon alfa-2b; Ribavirin; grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grazoprevir + Elbasvir (Experimental): Participants receive a fixed-dose combination (FDC) tablet of 100 mg grazoprevir and 50 mg elbasvir for 12 weeks, followed by 24 weeks of follow-up.
  Interventions: Drug: Sofosbuvir; Biological: PegIntron; Drug: Ribavirin
- SOF + PR (Active Comparator): Participants receive SOF (400 mg) combined with PegIntron (1.5 mcg/kg) plus RBV (1000-1200 mg weight-based dose) for 12 weeks, followed by 24 weeks of follow-up.
  Interventions: Drug: Grazoprevir/Elbasvir (100 mg/50 mg) FDC

INTERVENTIONS:
Drug: Sofosbuvir — 400 mg tablets, taken orally (PO) every day (QD) for 12 weeks.
  Arms: Grazoprevir + Elbasvir
Biological: PegIntron — PegIntron administered subcutaneously every week (QW) at 1.5 mcg/kg for 12 weeks.
  Arms: Grazoprevir + Elbasvir
Drug: Ribavirin — Capsule and/or tablet administered PO twice daily (BID) based on weight (1000 - 1200 mg) for 12 weeks.
  Arms: Grazoprevir + Elbasvir
Drug: Grazoprevir/Elbasvir (100 mg/50 mg) FDC — Grazoprevir/Elbasvir (100 mg/50 mg) FDC, taken PO QD for 12 weeks.
  Arms: SOF + PR

SUMMARY:
This is a study comparing grazoprevir (MK-5172) plus elbasvir (MK-8742) treatment with sofosbuvir (SOF) plus Pegylated Interferon plus Ribavirin (RBV) [PR] treatment in treatment-naïve and prior PR treatment failure participants with chronic Hepatitis C Virus (HCV) genotype (GT)1, GT4, or GT6 infection. The primary objectives are to compare efficacy (assessed by the percentage of participants achieving sustained virologic response 12 weeks after ending study treatment [SVR12]) and safety between the grazoprevir plus elbasvir treatment arm and the SOF plus PR treatment arm. The primary hypothesis is that the percentage of participants achieving SVR12 in the grazoprevir plus elbasvir treatment arm is non-inferior to that in the SOF plus PR treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Weigh ≥40 kg and ≤125 kg
* documented chronic HCV GT1, GT4, or GT6 infection
* cirrhosis/absence of cirrhosis defined by liver biopsy, Fibroscan, or FibroSure®
* either treatment naïve or PR Null Responder, PR Partial Responder, or PR Prior Relapser
* participant and partner both agree to use at least use at least 2 effective methods of contraception from at least 2 weeks prior to Day 1 and continue until up to 6 months after last dose of study drug, or longer if dictated by local regulations

Exclusion Criteria:

* has evidence of decompensated liver disease
* is coinfected with hepatitis B virus (e.g. hepatitis B surface antigen positive) or human immunodeficiency virus
* history of malignancy ≤5 years prior to signing informed consent, or is under evaluation for other active or suspected malignancy
* has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* has any of the following conditions: immunologically-mediated disease, organ transplants other than cornea and hair, poor venous access that precludes routine peripheral blood sampling, history of gastric surgery or malabsorption disorders, or any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial, history of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2015-11-26 (Actual); Study Completion 2016-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sperl J, Horvath G, Halota W, Ruiz-Tapiador JA, Streinu-Cercel A, Jancoriene L, Werling K, Kileng H, Koklu S, Gerstoft J, Urbanek P, Flisiak R, Leiva R, Kazenaite E, Prinzing R, Patel S, Qiu J, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Platt HL. Efficacy and safety of elbasvir/grazoprevir and sofosbuvir/pegylated interferon/ribavirin: A phase III randomized controlled trial. J Hepatol. 2016 Dec;65(6):1112-1119. doi: 10.1016/j.jhep.2016.07.050. Epub 2016 Aug 16. PMID 27542322
- [Derived] Ng X, Nwankwo C, Arduino JM, Corman S, Lasch KE, Lustrino JM, Patel S, Platt HL, Qiu J, Sperl J. Patient-reported outcomes in individuals with hepatitis C virus infection treated with elbasvir/grazoprevir. Patient Prefer Adherence. 2018 Dec 11;12:2631-2638. doi: 10.2147/PPA.S172732. eCollection 2018. PMID 30587935
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687
- [Derived] Reau N, Robertson MN, Feng HP, Caro L, Yeh WW, Nguyen BT, Wahl J, Barr E, Hwang P, Klopfer SO. Concomitant proton pump inhibitor use does not reduce the efficacy of elbasvir/grazoprevir: A pooled analysis of 1,322 patients with hepatitis C infection. Hepatol Commun. 2017 Aug 22;1(8):757-764. doi: 10.1002/hep4.1081. eCollection 2017 Oct. PMID 29404492
- [Derived] Zeuzem S, Serfaty L, Vierling J, Cheng W, George J, Sperl J, Strasser S, Kumada H, Hwang P, Robertson M, Wahl J, Barr E, Talwani R, Platt H. The safety and efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 1b infection. J Gastroenterol. 2018 May;53(5):679-688. doi: 10.1007/s00535-018-1429-3. Epub 2018 Jan 17. PMID 29344726

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 257 participants were randomized to treatment: 129 to Grazoprevir + Elbasvir arm and 128 to Sofosbuvir plus Pegylated Interferon/Ribavirin (SOF + PR) arm. Two participants in the SOF + PR arm withdrew from study prior to treatment.
Period: Overall Study
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Started | 129 | 128
Treated | 129 | 126
Completed | 127 (Completed = Completed Follow-up Week 24 (end of study)) | 121 (Completed = Completed Follow-up Week 24 (end of study))
Not Completed | 2 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS); all randomized participants who receive at least one dose of study treatment. Two participants in the SOF + PR arm withdrew from study prior to treatment and were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Grazoprevir + Elbasvir | SOF + PR | Total
Number analyzed (Participants) | 129 | 126 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.4) | 48.2 (12.4) | 47.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 64 | 138
  Male | 55 | 62 | 117

OUTCOME MEASURES:

1. Primary Outcome: Primary: Percentage of Participants Achieving Sustained Virologic Response at 12 Weeks After the End of All Treatment (SVR12)
Description: Hepatitis C Virus ribonucleic acid (HCV-RNA) levels in plasma were measured using the Roche COBAS®AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 on blood samples drawn from each participant. SVR12 was defined as HCV RNA below the lower limit of quantification (<LLOQ) at 12 weeks after the end of all study therapy. The primary efficacy hypothesis for this study was that the percentage of participants achieving SVR12 in the grazoprevir plus elbasvir arm was non-inferior to the percentage in the SOF plus PR arm. A secondary statistical analysis was performed to determine whether the percentage of participants achieving SVR12 in the grazoprevir plus elbasvir arm was superior to the percentage in the SOF plus PR arm.
Time Frame: 12 weeks after end of all therapy (Study Week 24)
Population: FAS; all randomized participants who receive at least one dose of study treatment. Two participants in the SOF + PR arm withdrew from study prior to treatment and were excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Number analyzed (Participants) | 129 | 126
percentage of participants | 99.2 | 90.5
Statistical Analysis 1: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Primary Analysis Approach: Non-Inferiority Analyses of the percentage of participants achieving SVR12 was conducted using the Miettinen & Nurminen (M&N) method. The analysis was adjusted for genotype (1a vs. non-1a) and fibrosis stage (cirrhotic vs. non-cirrhotic). The adjusted differences (grazoprevir+elbasvir arm minus SOF+PR arm) in percentages along with the corresponding 95% confidence intervals (CIs) and p-values were provided; Test type: Non-Inferiority or Equivalence — The lower bound of 95% CIs was compared to pre-specified non-inferiority margin, -10% to evaluate non-inferiority. The Missing=Failure (M=F) approach was used to handle missing values; p < 0.001, Miettinen & Nurminen Method; Adjusted Difference in Percentage = 8.8, 95% CI 2-sided [3.6 to 15.3]
Statistical Analysis 2: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Secondary Analysis Approach: Superiority Analyses of the percentage of participants achieving SVR12 was conducted using the M&N method. The analysis was adjusted for genotype (1a vs. non-1a) and fibrosis stage (cirrhotic vs. non-cirrhotic). The adjusted differences (grazoprevir +elbasvir arm minus SOF+PR arm) in percentages along with the corresponding 95% CIs and p-values were provided; Test type: Superiority or Other; p = 0.001, Miettinen & Nurminen Method; The lower bound of 95% CIs was compared to zero to evaluate superiority. The M=F approach was used to handle missing values; Adjusted Difference in Percentage = 8.8, 95% CI 2-sided [3.6 to 15.3]

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE) During the Treatment Period Plus First 14 Follow-up Days
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an AE. The percentage of participants who experienced at least one AE was reported for each treatment arm.
Time Frame: Treatment + First 14 days of follow-up (Up to Week 14)
Population: All Subjects as Treated (ASaT) population; all randomized participants who received at least one dose of study treatment. Two participants in the SOF + PR arm withdrew from study prior to treatment and were excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Number analyzed (Participants) | 129 | 126
percentage of participants | 51.9 | 93.7
Statistical Analysis 1: Comparison: Grazoprevir + Elbasvir vs SOF + PR; The percentage of participants with an event were assessed via point estimates with 95% CIs provided for between-group comparisons; Test type: Superiority or Other; Difference in Percentage = -41.7, 95% CI 2-sided [-51.1 to -31.9]

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an AE.
  The percentage of participants who discontinued study treatment due to an AE was reported for each treatment arm. Participants that discontinued study drug treatment due to an AE may have still continued on trial.
Time Frame: Up to Week 12
Population: ASaT population; all randomized participants who received at least one dose of study treatment. Two participants in the SOF + PR arm withdrew from study prior to treatment and were excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Number analyzed (Participants) | 129 | 126
percentage of participants | 0.8 | 0.8

4. Secondary Outcome: Percentage of Participants Experiencing at Least One Tier 1 Safety Event (Key Safety Parameter) During the Treatment Period and First 14 Follow-up Days
Description: Tier 1 safety events were pre-specified by the protocol to evaluate safety and test the safety superiority hypothesis. Tier 1 safety events were chosen to assess broad tolerability, hematological side effects and liver-related laboratory abnormalities. For this study, Tier 1 safety events included: any serious drug-related AE, any drug-related AE leading to permanent discontinuation (DC) of all study drugs, neutrophil count <0.75 x 10^9/L, hemoglobin <10 g/dL, severe depression, hepatic events of clinical interest (defined by abnormal increases in alanine aminotransferase [ALT], aspartate aminotransferase [AST], or alkaline phosphatase [ALP]), or events meeting stopping rule criteria for DC from trial (due to abnormal increases of ALT, AST, or ALP with/without pre-specified related AEs). The percentage of participants who experienced each individual event that was defined as a Tier 1 safety event during the study treatment period was reported for each treatment arm.
Time Frame: Treatment + First 14 days of follow-up (Up to Week 14)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Number analyzed (Participants) | 129 | 126
percentage of participants
  Total Tier 1 AEs | 0.8 | 27.8
  Tier 1 AE: Serious drug-related AE | 0.0 | 2.4
  Tier 1 AE: DC due to drug-related AE | 0.0 | 0.8
  Tier 1 AE: Neutrophil count <0.75 x 10^9/L | 0.0 | 12.7
  Tier 1 AE: Hemoglobin <10 g/dL | 0.8 | 14.3
  Tier 1 AE: Severe depression | 0.0 | 0.0
  Tier 1 AE: Hepatic event of clinical interest | 0.0 | 0.0
  Tier 1 AE: Trial DC due to stopping rule | 0.0 | 0.0
Statistical Analysis 1: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Total Tier 1 AEs: If, and only if the primary efficacy null hypothesis was rejected, the Tier 1 safety superiority hypothesis was tested at the 2-sided 5% alpha level. The safety superiority hypothesis was that the percentage of grazoprevir+elbasvir participants with ≥1 Tier 1 event is lower than the percentage of SOF+PR participants with ≥1 Tier 1 event; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen Method — % of participants with ≥1 Tier 1 event = total number participants with ≥1 Tier 1 event ÷ total number ASaT participants within each treatment arm. M&N method used to calculate a 2-sided 95% CI for the treatment difference and corresponding p-value; Difference in Percentage = -27.0, 95% CI 2-sided [-35.5 to -19.6]
Statistical Analysis 2: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Serious drug-related AEs: If, and only if the primary efficacy null hypothesis was rejected, the Tier 1 safety superiority hypothesis was tested at the 2-sided 5% alpha level. The safety superiority hypothesis was that the percentage of grazoprevir+elbasvir participants with ≥1 Tier 1 event is lower than the percentage of SOF+PR participants with ≥1 Tier 1 event; Test type: Superiority or Other; p = 0.078, Miettinen & Nurminen Method — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = -2.4, 95% CI 2-sided [-6.8 to 0.6]
Statistical Analysis 3: Comparison: Grazoprevir + Elbasvir vs SOF + PR; DC due to drug-related AE: If, and only if the primary efficacy null hypothesis was rejected, the Tier 1 safety superiority hypothesis was tested at the 2-sided 5% alpha level. The safety superiority hypothesis was that the percentage of grazoprevir+elbasvir participants with ≥1 Tier 1 event is lower than the percentage of SOF+PR participants with ≥1 Tier 1 event; Test type: Superiority or Other; p = 0.312, Miettinen & Nurminen Method — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = -0.8, 95% CI 2-sided [-4.4 to 2.1]
Statistical Analysis 4: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Neutrophil count <0.75 x 10^9/L: If, and only if the primary efficacy null hypothesis was rejected, the Tier 1 safety superiority hypothesis was tested at the 2-sided 5% alpha level. The safety superiority hypothesis was that the percentage of grazoprevir+elbasvir participants with ≥1 Tier 1 event is lower than the percentage of SOF+PR participants with ≥1 Tier 1 event; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen Method — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = -12.7, 95% CI 2-sided [-19.7 to -8.0]
Statistical Analysis 5: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Hemoglobin <10 g/dL: If, and only if the primary efficacy null hypothesis was rejected, the Tier 1 safety superiority hypothesis was tested at the 2-sided 5% alpha level. The safety superiority hypothesis was that the percentage of grazoprevir+elbasvir participants with ≥1 Tier 1 event is lower than the percentage of SOF+PR participants with ≥1 Tier 1 event; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen Method — [p-value comment as in outcome 4, analysis 1]; Difference in Percentage = -13.5, 95% CI 2-sided [-20.8 to -7.9]

5. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After Ending Study Treatment (SVR24)
Description: HCV-RNA levels in plasma were measured using the Roche COBAS®AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 on blood samples drawn from each participant. SVR24 was defined as HCV RNA <LLOQ at 24 weeks after the end of all study therapy.
Time Frame: 24 weeks after end of all therapy (Study Week 36)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Number analyzed (Participants) | 129 | 126
percentage of participants | 98.4 | 89.7
Statistical Analysis 1: Comparison: Grazoprevir + Elbasvir vs SOF + PR; Analyses of the percentage of participants achieving SVR24 was conducted using the Miettinen & Nurminen (M&N) method. The analysis was adjusted for genotype (1a vs. non-1a) and fibrosis stage (cirrhotic vs. non-cirrhotic). The adjusted differences (grazoprevir+elbasvir arm minus SOF+PR arm) in percentages along with the corresponding 95% confidence intervals (CIs) and p-values were provided; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Difference in Percentage = 8.8, 95% CI 2-sided [3.3 to 15.7]

6. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 4 Weeks After Ending Study Treatment (SVR4)
Description: HCV-RNA levels in plasma were measured using the Roche COBAS®AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 on blood samples drawn from each participant. SVR4 was defined as HCV RNA <LLOQ at 4 weeks after the end of all study therapy.
Time Frame: 4 weeks after end of all therapy (Study Week 16)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Number analyzed (Participants) | 129 | 126
percentage of participants | 99.2 [95.8 to 100.0] | 92.1 [85.9 to 96.1]

ADVERSE EVENTS:
Time Frame: Up to Follow-up Week 24
Description: ASaT population; all randomized participants who received at least one dose of study treatment. Two randomized participants in the SOF + PR arm withdrew from study prior to treatment and were excluded from analysis.
Arm/Group | Grazoprevir + Elbasvir | SOF + PR
Serious Adverse Events (participants affected / at risk) | 1/129 | 6/126
Other Adverse Events (participants affected / at risk) | 44/129 | 114/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir + Elbasvir (N=129) | SOF + PR (N=126)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Proctitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir + Elbasvir (N=129) | SOF + PR (N=126)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 15 (15)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 11 (15)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 8 (10)
Nausea (Gastrointestinal disorders) | 8 (9) | 13 (23)
Asthenia (General disorders) | 8 (10) | 30 (36)
Chills (General disorders) | 2 (4) | 21 (27)
Fatigue (General disorders) | 9 (9) | 32 (48)
Influenza like illness (General disorders) | 1 (1) | 23 (40)
Pyrexia (General disorders) | 2 (2) | 68 (191)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 8 (12)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 16 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 14 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 19 (47)
Dizziness (Nervous system disorders) | 4 (5) | 7 (10)
Headache (Nervous system disorders) | 17 (31) | 50 (97)
Irritability (Psychiatric disorders) | 0 (0) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (27)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.